CLINICAL TRIAL: NCT05513846
Title: Brain Age and Sleep Architecture in Meditators
Acronym: BRANCH
Status: Completed | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Balachundhar Subramaniam, Principal Investigator, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000597
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Brain Age

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Meditation: This is the group that will have learned at least Shamhbavi Mahamudra Kriya before they are enrolled in the study.
  Interventions: Device: DREEM EEG Device; Device: SleepImage Ring
- Control: This is the group that will not have learned Shambhavi Mahamudra Kriya before they are enrolled in the study. They will be invited to the study by the Meditation group.
  Interventions: Device: DREEM EEG Device; Device: SleepImage Ring

INTERVENTIONS:
Device: DREEM EEG Device — The DREEM EEG device will be used to measure brain age.
Device: SleepImage Ring — The SleepImage ring uses plethysmography to analyze sleep architecture and cardiopulmonary coupling.

SUMMARY:
This is a single-center, cross-sectional study that will recruit approximately fifty seven (57) meditators and fifty one (51) controls. Individuals that have learned at least the Shambhavi Mahamudra Kriya practice and live in Massachusetts will be mailed a DREEM EEG device, and a sleepimage ring. Participants will be asked to wear the two devices while sleeping for three consecutive weekday nights (Sunday night to Thursday night) and two weekend nights (Friday and Saturday nights). While meditating during the day, participants will only wear the DREEM EEG headband. Participants will also undergo neurocognitive tests from the NIH toolbox during one virtual visit via video call. Meditators who join the study will be asked to invite a control subject to the study, matched for age and comorbidities.

DETAILED DESCRIPTION:
Approximately one hundred and eight (108) individuals will undergo three consecutive weekday nights and two weekend nights of EEG and plethysmography recording using the DREEM headband and SleepImage rings, after answering a demographic questionnaire. Out of these 108 participants, the study will aim for 57 meditators and 51 matched controls. Only meditating participants will be asked to perform the most advanced form of meditation among the following three, which are listed from least advanced to most advanced: Shambhavi Mahamudra Kriya, Shoonya Meditation, Samyama Meditation (Breath watching). Participants will be instructed to wear the DREEM EEG headband during their practice of this meditation during each of the five days.

All participants will also be asked to undergo cognitive assessments from the NIH toolbox during a video call. The assessments from the NIH toolbox will last approximately forty-five minutes to one hour.

EEG: The participants will be mailed the DREEM devices and asked to wear them for three consecutive weekday nights and two weekend nights while sleeping. During the day, for each of these five nights, meditating participants will also be asked to wear the device while they sit still with their eyes closed, without trying to meditate, for 10 minutes. This will function as the baseline waking EEG measurement. Immediately following this, participants will be asked to perform their meditation while wearing the DREEM device for a maximum of 30 minutes.

NIH Toolbox:

This study will use select tests from the NIH Toolbox Cognition Battery and from the NIH Toolbox Emotion Battery. All of the tests together will take approximately 45 minutes to 1 hour to complete.

The selected tests from the batteries are the following:

Cognition Battery

1. Picture vocabulary test
2. List sorting working memory test
3. Picture Sequence Memory test
4. Oral reading recognition test

Emotion Battery:

1. Positive Affect CAT
2. General Life Satisfaction CAT
3. Emotional Support FF
4. Instrumental Support FF
5. Friendship FF
6. Loneliness FF
7. Perceived Stress FF

ELIGIBILITY:
Inclusion Criteria (Meditators):

1. Previous experience with learning Shambhavi Mahamudra Kriya
2. Age 18 years or older.
3. Lives in the United States barring California

Inclusion Criteria (Controls):

1. Age 18 years or older
2. Lives in the United States barring California

Exclusion Criteria (both groups):

1. Non-English Speaking
2. Night Shift workers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will not be recruited based on race, ethnicity, or gender. However, it is not clear whether the final study sample will contain a representative spread of the racial and gender makeup.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-07-04 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Brain Age | Measured for 3 weekday and 3 weekend nights during the data collection period
  Brain Age will be calculated using an algorithm from the sleeping EEG. A Brain Age index score will be created for each participant based on an aggregate of the five days of sleeping EEG data. The Brain Age Index is the brain age calculated from the algorithm subtracted by the chronological age of the participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Centre, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No